

| Document Title: | Statistical Analysis Plan BIO CONCEPT.Renamic Neo |
|---|---|
| Document Version and Date: | Version 2-0, 18-Sep-2020 |
| ClinicalTrials.gov Identifier: | NCT04350008 |

Rev. B

| Sponsor: | BIOTRONIK Australia Pty. Ltd. |
|---|---|
| Study name / EAC code: | BIO Concept. Renamic Neo |
| Version and date of the Statistical Analysis Plan: | 2-0 from 18Sep2020 |
| Version and date of the underlying Clinical Investigation Plan: | 1-0 from 05Dec2019 |

| Print Name & Title | Signature | Date of Signature |
|---|---|---|
| | | (DD MMM YYYY) |
| Project Manager | | |
| BIOTRONIK SE & Co. KG Center for Clinical Research Woermannkehre 1 12359 Berlin | | |
| Germany | | |
| Scientist | | |
| BIOTRONIK SE & Co. KG Center for Clinical Research Woermannkehre 1 12359 Berlin | | |
| Germany | | |
| Biostatistician | | |
| BIOTRONIK SE & Co. KG<br>Center for Clinical Research<br>Woermannkehre 1<br>12359 Berlin | | |
| Germany | | |

# **Table of Content**

| Table of Content | 2 |
|----------------------------------------------------------------|----------|
| 0. Change History | 4 |
| 1. Introduction | 5 |
| 1.1. Aim | 5 |
| 1.2. General information | 5 |
| 2. Objectives | 7 |
| 3. Investigational Device | 7 |
| 4. Study Design & Time Course | 7 |
| 5. General Statistical Procedures | 9 |
| 5.1. Descriptive analyses | 9 |
| Nominal – dichotomous data | 9 |
| Nominal data – more than two categories | |
| Scale / metric data | 10 |
| Ordinal data | 10 |
| 5.2. Inferential analyses | 11 |
| 5.3. Significance level | 11 |
| 5.4. Missing Data | 11 |
| 5.5. Exclusion of data from confirmatory data analysis | 11 |
| 5.6. Subgroups | 11 |
| 5.7. Interim analyses | 11 |
| 5.8. Software | 11 |
| 5.9. CDMS export | 12 |
| Datasets to be analyzed based on this SAP Other Datasets | 12 |
| | 12 |
| 6. Specific Study Dates 6.1. Enrollment date | 13 |
| | 13<br>13 |
| <ul><li>6.2. Implantation date</li><li>6.1. PHD date</li></ul> | 13 |
| 6.1. FU date | 13 |
| 6.2. Termination date | 13 |
| 7. Analysis Sets & Subgroups | 14 |
| 7.1. Analysis Sets | 14 |
| Subgroups | 15 |
| 8. Data for a CONSORT diagram and "study realization" | 16 |
| 8.1. Analysis set | 16 |
| 8.2. Enrollment | 16 |
| Inclusion criteria | 16 |
| Exclusion criteria | 16 |
| 8.3. Termination | 17 |
| 8.4. Fu duration | 17 |
| 8.5. Investigations | 18 |
| 9. Baseline | 19 |
| 9.1. Analysis set | 19 |
| 9.2. Variables | 19 |
| Baseline / Demographic data | 19 |
| Medical history / Heart Failure | 19 |
| Medical history / Coronary Artery Disease | 19 |
| Medical history / Brady- and Tachyarrhythmias | 20 |
| Medical history / known comorbidities | 20 |
| 9.3. Treatment of Missing and Spurious Data | 21 |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



# Statistical Analysis Plan

| BIO | Concept. | Renamic | Neo | Version | 2-0 |
|-----|----------|---------|-----|---------|-----|

Page 3/48

| 9.4. Exclusion of Particular Information | | 21 |
|---|---|---|
| 9.5. Descriptive Analyses | | 21 |
| 9.6. Hypotheses & Statistical Tests | | 21 |
| 10. ADE and DD Endpoints - Implantatio | n | 22 |
| 10.1. Analysis Set and Data Selection | | 22 |
| 10.2. Variables | | 22 |
| Adjudicated Adverse Device Effects / Dev | | 22 |
| 10.3. Treatment of Missing and Spurio | | 24 |
| 10.4. Exclusion of Particular Information | on | 24 |
| 10.5. Descriptive Analyses | | 24 |
| 10.6. Hypotheses & Statistical Tests | | 24 |
| <ol> <li>ADE and DD Endpoints – PHD &amp; follo</li> </ol> | w-up | 25 |
| 11.1. Analysis Set and Data Selection | | 25 |
| 12. Implantation & PSA | | 26 |
| 12.1. Analysis Set | | 26 |
| 12.2. Variables | | 26 |
| Used Programmer Features: Pacing Sys | , , , | 26 |
| Used Measurement Mode: Pacing Syste | , , , | 27 |
| 12.1. Treatment of Missing and Spurio | | 28 |
| 12.2. Exclusion of Particular Information | on | 28 |
| 12.3. Descriptive Analyses | | 28 |
| 12.4. Hypotheses & Statistical Tests | | 28 |
| 13. General Assessments - Implantation | | 29 |
| 13.1. Analysis Set and Data Selection | | 29 |
| Used Programmer Features: Implant | | 30 |
| Accuracy of PSA Measurements | | 32 |
| Used Programmer Features: Data expo | rt | 33 |
| Used Programmer Features: Printing | | 34 |
| Used Programmer Features: Battery | | 34 |
| Assessment of Programmer Features | | 35 |
| 13.1. Treatment of Missing and Spurio | | 36 |
| 13.2. Exclusion of Particular Information | on | 36 |
| 13.3. Descriptive Analyses | | 36 |
| 13.4. Hypotheses & Statistical Tests | | 36 |
| 14. General Assessments – PHD & Follow | <i>ı-</i> up | 37 |
| 14.1. Analysis Set and Data Selection | | 37 |
| 15. Devices and Accessories - Implantation | on | 38 |
| 15.1. Analysis Set and Data Selection | | 38 |
| Implanted Devices | | 38 |
| Renamic Neo and software | | 39 |
| ECG cable | | 40 |
| Electrode clip | | 41 |
| Patient cable | | 42 |
| Patient adapter | | 44 |
| Accessory bag | | 45 |
| 15.2. Treatment of Missing and Spurio | | 46 |
| 15.3. Exclusion of Particular Information | วท | 46 |
| 15.4. Descriptive Analyses | | 46 |
| 15.5. Hypotheses & Statistical Tests | | 46 |
| 16. Devices and Accessories – PHD & following | ow-up | 47 |
| 16.1. Analysis Set and Data Selection | | 47 |



# 0. Change History

Version 1.0: Initial document.

Version 2-0: Final version before CDMS-freeze for interim analysis; implementation of new internal adjudication dataset;

implementation of findings during blind review (spurious implantation date);

routine document improvements and corrections.



# 1. Introduction

#### 1.1. Aim

The aim of this document is to provide detailed instructions on all descriptive and inferential statistical analyses for the Clinical Investigation Report (CIR). Inferential analyses of the primary and secondary endpoint(s) as defined in this document are mandatory to be reported in the CIR.

#### 1.2. General information

The text contains verbatim excerpts from the CIP. Such excerpts are italicized with grey background; e.g.

....

The main aspects and the design of the clinical investigation are presented in chapters 1-4.

General statistical procedures are summarized in chapter 5. Those methods are used in case there is no other specification within this document.

Definitions of the specific dates, e.g. enrollment and termination are presented in chapter 6.

Specific analysis sets are defined in chapter 7.

Descriptive and inferential statistical analyses are handled in following chapters.

Thereby the following statistical considerations are specified:

- Definition of the analysis set for the following analyses, e.g. excluding patients without any measured or imputed data for this endpoint.
- Definition of the endpoint(s) to be analyzed including references to the source data, e.g. CRF sheet and item.
- Treatment of missing and spurious data for evaluation of the above endpoint(s).
- Exclusion of particular information from the evaluation of the above endpoint(s) in addition to the exclusion of patients from the analysis set.
- Descriptive analyses including tables and figures
- Statistical alternative hypothesis/hypotheses (HA) to analyze the above endpoint(s) if available.
- Statistical tests intended to analyze the above hypothesis/hypotheses if available.



All variables are defined in tables using the following columns:

Data file
 Name of a data file exported from the CDMS with one data row per unique identifier (e.g. patient-specific "patient display ID full" or event-specific record ID); additionally, a new data file ("data SAR") might be generated by merging all relevant data from the original CDMS data files and generating derived variables (e.g. BMI from weight and height or date

of first AE episode)

Notes Information whether data has to be presented with

"descriptive" methods as defined in the following sub-chapter, data for "case listings" of original data for each patient specified, or "no report" for data needed for generating of derived variables only

• Variable name Original name of a variable in the CDMS data file or

name of a derived variables (indicated with a suffix "SAR");

Variable label
 Original labels from the CDMS data will be used for generating the SAR

unless a new label is defined in this document ("NEW"); labels might be omitted or shortened ("...") if remaining clear

Variable level Nominal, ordinal, scale (metric, continuous), or date

Nominal values
 Original values from CDMS data will be used for generating the SAR

unless new nominal values are defined in this document ("NEW"); values might be omitted or shortened ("...") if remaining clear;

for numeric data this information is not applicable (n.a.)

| Data file, identifier | Notes | Variable | Variable | Variable | Nominal |
|-------------------------|-------|----------|----------|----------|---------|
| patient display id full | | name | label | level | values |



# 2. Objectives

### CIP chapter 7.1 Objectives

This study is designed as a pre-market clinical study to provide evidence on the safety, performance and usability of the Renamic Neo programmer hardware, software and ECG cable PK-222-L to support regulatory approval, with a focus on requirements of the European Medical Device Regulation (MDR). The study is also intended to identify and evaluate residual risks associated with the use of the Renamic Neo programmer system that remained unrevealed even after risk analysis, risk mitigation and completed validation of the device. The results will be used to update the clinical evaluation of the devices.

# 3. Investigational Device

### CIP chapter 4.7.1 Renamic Neo hardware and software

The Renamic Neo programmer system comprises the Renamic Neo hardware, software and the ECG cable PK-222-L. The functional design is highly similar to the predecessor Renamic. Some software features related to PSA functionalities and the graphical user interface (GUI) have been optimized and are described below. The hardware consists of the Renamic Neo, the programmer head (PGH), the battery and the pacing system analyzer (PSA). Several accessories can be used with the programmer to record ECG or to conduct lead positioning checks during implantations. These include ECG cables, patient cables, electrode clips and patient adapters.

...

# 4. Study Design & Time Course

#### CIP chapter

Patients will be enrolled either for implantation including subsequent pre-hospital discharge or for a follow-up visit only. ICM patients will be included for follow-ups only. As the total study duration is planned for only 3 months different patients will be included for implantation and for follow-up. Patients that have been enrolled in the study and were terminated shall not be included a second time in the study.

...



Table 3: Overview of study procedures

| Investigations | Enrollment /<br>Baseline | For patients enrolled before implantation | | For patients<br>enrolled after<br>implantation |
|---|---|---|---|---|
| | | Implantation | Pre-hospital<br>discharge | Follow-up |
| Patient informed consent | x | | | |
| Verification of in- and exclusion criteria | × | | | |
| Demographics and medical history | x | | | |
| Information on implanted IPG, ICD,<br>CRT or ICM, leads (device log) | x* | x | | |
| PSA measurements and evaluation | | × | | |
| Device based measurements and evaluation, if applicable | | x | x | × |
| Evaluation of implant interrogation and programming functionality | | х | х | x |
| General assessment of Renamic Neo<br>hardware and software | | x | x | × |
| Evaluation of usability of Renamic Neo system | | X | х | × |
| Data export (connectivity, printing) | | x | х | x |
| Data export of use case data for<br>evaluation at sponsor | | x | x | × |
| Used accessories (including entry in device log) | | х | х | × |
| Battery usage | | × | × | × |
| Adverse event and device deficiency reporting | × | × | × | × |
| Concomitant medication | x <sup>1</sup> | x <sup>1</sup> | x <sup>1</sup> | x <sup>1</sup> |
| Regular termination | | | х | x |

x point in time of study procedure depends if patient is enrolled for implantation use case (includes PHD) or for follow-up use case.



x\* point in time for follow-up cases

x1 only if related to an AE

# 5. General Statistical Procedures

# 5.1. Descriptive analyses

# CIP chapter 11.1 Statistical design, method and analytical procedures

For continuous variables descriptive statistics (mean, standard deviation, median, quartiles, minimum, and maximum) will be calculated. For nominal and ordinal variables absolute and relative frequencies will be calculated based on non-missing data. Ordinal variables are described similar as continuous data (minimum, median, quartiles, and maximum) or by absolute and relative frequencies based on non-missing data of each category. Further details will be provided in the separate Statistical Analysis Plan (SAP).

For illustration, see the following standard tables with and without subgroup analyses based on dummy data.

### Nominal - dichotomous data

| | | | | Relative |
|--------------------------------|----------|---------|-----------|-----------|
| Variable | | N non- | Absolute | frequency |
| (N total = 10) | Category | missing | frequency | [%] |
| Gender | Female | 9 | 3 | 33.3 |
| History of atrial fibrillation | Yes | 8 | 4 | 50.0 |

| | | | | | Relative |
|---|---|---|---|---|---|
| Variable | | Group | N non- | Absolute | frequency |
| (N total = 10) | Category | Type of implanted device | missing | frequency | [%] |
| Gender Female | | ICD (N group = 4) | 4 | 1 | 25.0 |
| | | CRT (N group = 4) | 4 | 2 | 50.0 |
| | | All | 9 | 3 | 33.3 |
| History of atrial fibrillation | Yes | ICD | 4 | 2 | 50.0 |
| | | CRT | 4 | 2 | 50.0 |
| | | All | 8 | 4 | 50.0 |

### Nominal data - more than two categories

| Variable | N non- | I | II | II | IV |
|----------------|---------|-----------|-----------|-----------|-----------|
| (N total = 10) | missing | N(%) | N(%) | N(%) | N(%) |
| NYHA class | 8 | 1 (12.5%) | 3 (37.5%) | 3 (37.5%) | 1 (12.5%) |

| Variable<br>(N total = 10) | Group Type of implanted device | N non-<br>missing | I<br>N(%) | II<br>N(%) | II<br>N(%) | IV<br>N(%) |
|---|---|---|---|---|---|---|
| NYHA Class | ICD (N group = 4) | 3 | 0 (0.0%) | 1 (33.3%) | 2 (66.7%) | |
| | CRT (N group = 4) | 4 | 1 (25.0%) | 1 (25.0%) | 1 (25.0%) | 1 (25.0%) |
| | All | 8 | 1 (12.5%) | 3 (37.5%) | 3 (37.5%) | 1 (12.5%) |



# Scale / metric data

| Variable | N non- | | | | Lower | | Upper | |
|---|---|---|---|---|---|---|---|---|
| (N total = 10) | missing | Mean | SD | Min | quartile | Median | quartile | Max |
| Age [years] | 9 | 56.1 | 15.9 | 25.0 | 50.0 | 60.0 | 66.0 | 77.0 |
| Weight [kg] | 8 | 78.5 | 13.9 | 55.0 | 69.5 | 78.5 | 89.0 | 99.0 |

| Variable | Group Type of implanted | N non- | | | | Lower | | Upper | |
|---|---|---|---|---|---|---|---|---|---|
| (N total = 10) | device | missing | Mean | SD | Min | quartile | Median | quartile | Max |
| Age [years] | ICD (N group = 4) | 4 | 61.8 | 11.2 | 50.0 | 55.0 | 60.0 | 68.5 | 77.0 |
| | CRT (N group = 4) | 4 | 50.3 | 21.5 | 25.0 | 32.5 | 53.0 | 68.0 | 70.0 |
| | All | 9 | 56.1 | 15.9 | 25.0 | 50.0 | 60.0 | 66.0 | 77.0 |
| Weight [kg] | ICD | 3 | 85.0 | 7.0 | 77.0 | 77.0 | 88.0 | 90.0 | 90.0 |
| | CRT | 4 | 76.0 | 18.5 | 55.0 | 62.5 | 75.0 | 89.5 | 99.0 |
| | All | 8 | 78.5 | 13.9 | 55.0 | 69.5 | 78.5 | 89.0 | 99.0 |

# Ordinal data

Identical tables as for metric data but without mean and SD



# 5.2. Inferential analyses

CIP chapter 11.3 Level of significance and the power of the study

Because there are no pre-specified hypotheses, all analyses will be exploratory.

...

### 5.3. Significance level

### CIP chapter 11.3 Level of significance and the power of the study

Because there are no pre-specified hypotheses, all analyses will be exploratory. For inferential analyses, a two-sided p-value less than 5% will be considered statistically significant. In accordance to the exploratory approach there will be no adjustment for multiplicity.

...

# 5.4. Missing Data

### CIP chapter 11.11 Handling of missing, unused and spurious data

For the endpoints, missing data will not be imputed.

Free text will be used to clarify other data.

Spurious data will be clarified via the query management system, i.e. corrected after approval of an investigator. Remaining outliers will be identified during the review of the data before CDMS closure. In case of a clear evidence of a measurement error, the Statistical Analysis Plan will be updated in order to avoid any bias. Spurious data, which were not clarified by the query process before CDMS freeze or closure, will be indicated. If appropriate, analyses will be performed both with/without such data.

# 5.5. Exclusion of data from confirmatory data analysis

# CIP chapter 11.12 Exclusion of data from the confirmatory data analysis

No data are documented or analyzed from patients without documented informed consent.

# 5.6. Subgroups

#### CIP chapter 11.9 Specification of subgroups

Potential critical events will be analyzed whether there is any connection to the subgroups IPG, ICD, CRT, or ICM.

#### 5.7. Interim analyses

### CIP chapter 11.6 Provision for an interim analysis

There is one planned interim analyses for internal purposes. Except for safety reasons no investigator is informed about the results and, thus, no bias is expected. There will be no adjustment for multiplicity.

### 5.8. Software

All analyses will be carried out using validated software, e.g. SAS version 9.4 or upgrades.



# 5.9. CDMS export

### Datasets to be analyzed based on this SAP

| Dataset<br>name | Data rows,<br>unique identifier<br>variables except record id | Data rows<br>unique identifier<br>description | Parent CRF<br>In case of<br>embedded<br>log | Notes |
|---|---|---|---|---|
| enrollment | patient display id full | Patient | n.a. | |
| baseline | patient display id full | Patient | n.a. | |
| Medical history | patient display id full | Patient | n.a. | |
| implantation<br>psa | patient display id full | Patient | n.a. | |
| general<br>assessments | patient display id full & autom SVTYP | Patient & visit type | n.a. | Visit type:<br>Implantation,<br>pre-hospital discharge follow-up (PHD),<br>regular follow-up after PHD |
| accessory<br>log details | patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | Patient & visit type & model & programmer serial no. | n.a. | Accessories: Renamic Neo programmer, ECG cable, electrode clip, patient cable, patient adapter |
| device log<br>details | patient display id full & DIDVTYP | Patient &<br>device type | n.a. | Device type: Pacemaker (single/dual chamber), ICD (single/dual chamber) CRT-P device, CRT-D device, ICM (Insertable Cardiac Monitor) RA lead, RV lead LV lead, VCS lead |
| adverse<br>event | n.a. | Event | n.a. | |
| internal<br>adjudication | n.a. | Event | n.a. | |
| device<br>deficiency | n.a. | Event | n.a. | Investigational device:<br>Renamic Neo Programmer,<br>Renamic Neo Programmer Software,<br>PK-222-L ECG cable |
| study<br>termination | patient display id full | Patient | n.a. | |

# Other Datasets

| Dataset<br>name | Data rows,<br>unique identifier<br>variables except record id | Data rows<br>unique identifier<br>description | Parent CRF<br>in case of<br>embedded<br>log | Notes |
|---|---|---|---|---|
| hospitalization<br>log | n.a. | Event | adverse<br>event | |
| device | DIDVTYP &<br>DIDVSNR | Device type &<br>device SNR / ID | n.a. | |
| deviation patient related | DVSPID | Deviation ID | n.a. | |
| deviation site related | DVSPID | Deviation ID | n.a. | |
| deviation<br>third party | DVSPID | Deviation ID | n.a. | |
| medication | patient display id full & CMTRT & CMSTDT | Patient & trade name & start date | n.a. | Documented in case of an adverse event. |





# 6. Specific Study Dates

### 6.1. Enrollment date

### CIP chapter 8.3.6 Point of enrollment and study termination

Point of enrollment is the date of signature of the informed consent form by the patient.

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient display id full | name | label | level | values |
| enrollment | DMICDT i | Patient dated ICF | date | n.a. |
| data SAR | date enr SAR = DMICDT i | Patient dated ICF | date | n.a. |

# 6.2. Implantation date

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient display id full | name | label | level | values |
| Implantation psa | PRIMSTDT i | Date of implantation | date | n.a. |
| baseline | SVSTDT_i | Date of baseline assessment | date | n.a. |
| data SAR | date imp SAR¹ | Date of implantation (excluding | date | n.a. |
| | | spurious data) | | |

#### 6.1. PHD date

| | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|
| for selection autom SVTYP = | SVFUSTDT i | Date of follow-up | date | n.a. |
| Pre-hospital discharge follow-up (PHD) | | | | |

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient display id full | name | label | level | values |
| data SAR | date PHD SAR = SVFUSTDT i | Date of PHD | date | n.a. |

### 6.1. FU date

| | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|
| general assessments | SVFUSTDT | Date of follow-up | date | n.a. |
| for selection autom SVTYP = | | | | |
| Regular follow-up after PHD | | | | |

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient display id full | name | label | level | values |
| data SAR | date FUP SAR = SVFUSTDT i | Date of regular follow-up | date | n.a. |
| | | after PHD | | |

### 6.2. Termination date

# CIP chapter 8.3.6 Point of enrollment and study termination

Date of regular termination for each patient is the date of discharge from the index hospitalization for implantation cases or the date of follow-up after follow-up completion for follow-up cases.

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| | | label | level | values |
| study termination | DSTRDT | Date of termination | date | n.a. |
| data SAR | Date ter SAR = DSTRDT i | Date of termination | date | n.a. |

 $<sup>^{1}</sup>$  IF PRIMSTDT i  $\geq$  SVSTDT\_i THEN date imp SAR $^{1}$  = PRIMSTDT i ELSE date imp SAR -> missing





#### **Analysis Sets & Subgroups** 7.

# 7.1. Analysis Sets

| Data file, identifier | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|
| patient display id full | name | label | level | |
| enrollment | DMSUBSPS | Patient signed the informed | nominal | o Yes |
| | | consent personally | | o No |
| enrollment | DMRPRSPS | An independent witness signed | nominal | ∘ Yes |
| | | the informed consent since the | | o No |
| | | patient is unable to write | | |
| study termination | DSDRPPRO | Please specify | nominal | <ul> <li>No implantation of an active</li> </ul> |
| | | Drop-out according to protocol | | implantable BIOTRONIK device |
| | | | | o Other |

| Data file, identifier patient display id full & autom SVTYP | | | Variable<br>level | Nominal values |
|---|---|---|---|---|
| general assessments | autom SVTYP | Visit type | | o Implantation<br>o Pre-hospital discharge follow-up (PHD)<br>o Regular follow-up after PHD |
| | | Was the Renamic Neo programmer used for the visit | nominal | o Yes<br>o No |

| Data file, identifier | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| patient display id full | name | label | level | values |
| data SAR | analysis set enr SAR <sup>2</sup> | Enrollment analysis set (patients with Biotronik | nominal | o Yes |
| | | device and usage of Renamic Neo) | | o No |
| data SAR | analysis set imp SAR <sup>3</sup> | Implantation analysis set (patients with Biotronik | nominal | o Yes |
| | | device and usage of Renamic Neo during implantation) | | o No |
| data SAR | analysis set PHD FUP SAR | PHD and regular FU analysis set (patients with | nominal | o Yes |
| | | Biotronik device and usage of Renamic Neo during PHD or FU) | | o No |

The implantation analysis set and the PHD/FUP analysis set are not mutually exclusive, i.e. specific patients can belong to both analysis sets.

THEN analysis set enr SAR = Yes ELSE analysis set enr SAR = No

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



<sup>&</sup>lt;sup>2</sup> IF (DMSUBSPS = Yes OR DMRPRSPS = Yes) AND date enr SAR not missing AND TIINC01 type ≠ No implantation of an active implantable BIOTRONIK device AND any general assessments per patient with PRSVPRG = Yes

<sup>3</sup> IF analysis set enr SAR = Yes AND

any general assessments per patient with (PRSVPRG = Yes AND autom SVTYP per patient = Implantation)

THEN analysis set imp SAR = Yes ELSE analysis set imp SAR = No

<sup>4</sup> IF analysis set enr SAR = Yes AND

any general assessments per patient with

<sup>([</sup>PRSVPRG = Yes AND autom SVTYP = Pre-hospital discharge follow-up (PHD)] OR

<sup>[</sup>PRSVPRG = Yes AND autom SVTYP = Regular follow-up after PHD])

THEN analysis set FUP SAR = Yes

ELSE analysis set FUP SAR = No

# Subgroups

| Data file, identifier patient display id full & DIDVTYP | | | Variable<br>level | Nominal values |
|---|---|---|---|---|
| device log details | 7,7 | hidden technical field: Short<br>name for<br>General type of device | | o CRT<br>o CRT-P<br>o ICD<br>o ICM<br>o IPG |

| Data file, identifier | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|
| patient display id full | name | label | level | |
| data SAR | subgroup device type SAR <sup>5</sup> | Subgroup type of device | nominal | o CRT |
| | | | | o CRT-P |
| | | | | o ICD |
| | | | | o ICM |
| | | | | o IPG |

<sup>&</sup>lt;sup>5</sup> Patient-specific type of device data for helpvar device type not missing subgroup device type SAR = helpvar device type



# 8. Data for a CONSORT diagram and "study realization"

# 8.1. Analysis set

Unless otherwise specified, all analyses are performed for the enrollment analysis set<sup>6</sup>.

### 8.2. Enrollment

- Date of FPI
- Date of LPI
- Number of patients
- Number of patients per site

### Inclusion criteria

| Data file,<br>identifier<br>patient<br>display id full | Notes | Variable<br>name | Variable<br>label | Variable<br>Ievel | Nominal values |
|---|---|---|---|---|---|
| enrollment | descri<br>ptive | | already has a BIOTRONIK active, implantable device | nominal | o Yes<br>o No |
| | | | Patient is able to understand the nature of<br>the study and provides written informed<br>consent | nominal | o Yes<br>o No |
| | | TIINC01<br>type | Type of inclusion criterion | nominal | o Patient is planned for de<br>novo implantation<br>o Patient has already an<br>implanted device |

# Exclusion criteria

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient | | | | | |
| display id full | | | | | |
| enrollment | descri | TIEXC01 | Patient is implanted with a Stratos pacemaker | nominal | ∘ Yes ∘ No |
| | ptive | TIEXC02 | Patient is pregnant or breastfeeding | nominal | ∘ Yes ∘ No |
| | | TIEXC03 | Patient is less than 18 years old | nominal | ∘ Yes ∘ No |
| | | TIEXC04 | Patient is planned for implant exchange or upgrade | nominal | ∘ Yes ∘ No |



<sup>&</sup>lt;sup>6</sup> analysis set enr SAR = Yes

### 8.3. Termination

- Date of FPO
- Date of LPO

| Data file:<br>Identifier<br>patient display<br>id full | | Variable<br>name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| termination | descriptive | DSRTRM | Regular study termination | 1 | o Yes<br>o No |
| | Descriptive for<br>DSRTRM = No | _ | Reason for<br>early study<br>termination | | o Patient moved away from investigational center o Patient is lost to follow-up o Patient withdrew consent to study participation o Patient death o Drop-out according to protocol o Enrollment failure |

| Data file:<br>Identifier<br>patient display<br>id full | Notes | Variable<br>name | Variable<br>label | Variable<br>Ievel | Nominal values |
|---|---|---|---|---|---|
| enrollment | Case case<br>listing for<br>DSETRREA = | DMICDT i | Patient: Date of<br>informed consent<br>signature | date | n.a. |
| | Drop-out<br>according to | DSTRDT i | Date of study<br>termination | date | n.a. |
| | protocol | DSDRPPRO | Reason for early study termination | nominal | o No implantation of an active implantable<br>BIOTRONIK device<br>o Other |
| | | CODRPPRO | Please specify<br>Drop-out according to<br>protocol - Other | text | |

# 8.4. Fu duration

The FU duration has to be analyzed separately for the implantation<sup>7</sup> and follow-up analysis set<sup>8</sup>.

| Data file:<br>Identifier | | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|
| patient display<br>id full | | | | |
| | descriptive and<br>cumulative sum | Days from enrollment to termination | scale | n.a |

<sup>9</sup> FU duration SAR = DSTRDT - DMICDT





<sup>&</sup>lt;sup>7</sup> analysis set imp SAR = Yes

 $<sup>^{8}</sup>$  analysis set FUP SAR = Yes

# 8.5. Investigations

The following frequency has to be analyzed for the implantation analysis set <sup>10</sup>.

| Data file:<br>Identifier<br>patient display<br>id full | | Variable<br>name | | <br>Nominal<br>values |
|---|---|---|---|---|
| data SAR | descriptive | PHD renamicneo SAR <sup>11</sup> | PHD with Renamic Neo | o Yes<br>o No |

The following frequencies have to be analyzed for the PHD/FUP analysis set12

| Data file: | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| Identifier | | name | label | level | values |
| patient display | | | | | |
| id full | | | | | |
| data SAR | descriptive | PHD renamicneo SAR | PHD with Renamic Neo | nominal | o Yes |
| | | | | | o No |
| data SAR | descriptive | FU renamicneo SAR <sup>13</sup> | Fu with Renamic Neo | nominal | o Yes |
| | | | | | o No |

<sup>&</sup>lt;sup>13</sup> If any general assessments per patient with (PRSVPRG = Yes AND autom SVTYP per patient = Regular follow-up after PHD) THEN PHD renamicneo SAR = Yes ELSE PHD renamicneo SAR = No





<sup>&</sup>lt;sup>10</sup> analysis set imp SAR = Yes

any general assessments per patient with

(PRSVPRG = Yes AND autom SVTYP per patient = Pre-hospital discharge follow-up (PHD))

THEN PHD renamicneo SAR = Yes

ELSE PHD renamicneo SAR = No

<sup>12</sup> analysis set PHD FUP SAR = Yes

# 9. Baseline

### CIP chapter 11.12 chapter 7.5 Further data of interest

General information

• Patient demographics and medical history

### 9.1. Analysis set

All analyses are performed for enrollment analysis set14.

#### 9.2. Variables

# Baseline / Demographic data

| Data file,<br>identifier patient<br>display id full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| baseline | descriptive | DMSEX | Gender | nominal | o Male<br>o Female |
| | descriptive | DMAGE | Age [Years] | scale | n.a. |
| baseline | descriptive | VSHGHT | Height [cm] | scale | n.a. |
| | descriptive | VSWGHT | Weight [kg] | scale | n.a. |
| | descriptive | VSBMI | BMI [kg/m2] | scale | n.a. |

### Medical history / Heart Failure

| Data file,<br>identifier patient<br>display id full | Notes | | | | Nominal<br>values |
|---|---|---|---|---|---|
| medical history | descriptive | MHHF | History of Heart failure | | ∘ Yes<br>∘ No |
| | descriptive for<br>MHHF = Yes | CVNYHA | | reported as nominal | 01<br>02<br>03<br>04 |

### Medical history / Coronary Artery Disease

| Data file,<br>identifier patient<br>display id full | Notes | | Variable<br>label | <br>Nominal<br>values |
|---|---|---|---|---|
| medical history | descriptive | MHCAD | History of coronary artery disease | <br><ul><li>Yes</li><li>No</li></ul> |
| | Descriptive for<br>MHCAD=Yes | MHMI | Prior myocardial infarction | <br>∘ Yes<br>∘ No |
| | | PRRVC | Prior revascularization (PCI or CABG) | <br>∘ Yes<br>∘ No |

<sup>&</sup>lt;sup>14</sup> analysis set enr SAR = Yes





# Medical history / Brady- and Tachyarrhythmias

| Data file,<br>identifier patient<br>display id full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| medical history | descriptive | MHSSS | History of sick sinus syndrome | nominal | o Yes<br>o No |
| | descriptive | MHAVB | History of AV block | nominal | o Yes<br>o No |
| | descriptive for<br>MHAVB =Yes | MHAVBTYP | Type of AV block | to be<br>reported as<br>nominal<br>variable | o1<br>o2<br>o3 |
| | descriptive | MHBBB | History of bundle branch block | nominal | ∘ Yes<br>∘ No |
| | descriptive | MHAFB | History of atrial fibrillation | nominal | ∘ Yes<br>∘ No |
| | descriptive for<br>MHAFB = Yes | CVAFBTYP | Type of atrial fibrillation | nominal | o Paroxysmal o Persistent o Long-standing persistent o Permanent |
| | descriptive | MHAVA | History of other<br>atrial/supraventricular<br>arrhythmias | nominal | o Yes<br>o No |
| | descriptive | MHVA | History of ventricular arrhythmias | nominal | o Yes<br>o No |

| Data file,<br>identifier patient<br>display id full | | | | | Nominal<br>values |
|---|---|---|---|---|---|
| imedical history | case listing for<br>MHAVA = Yes | | Specification of other type of atrial/supraventricular tachycardia | text | |
| | case listing for<br>MHVA = Yes | COAV | Specification of ventricular arrhythmias | text | |

# Medical history / known comorbidities

| Data file,<br>identifier patient<br>display id full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| medical history | descriptive | MHHP | Hypertension (including well-controlled) | nominal | ∘ Yes ∘ No |
| medical miscory | descriptive | MHVHD | Valvular heart disease | nominal | <ul><li>Yes ○ No</li></ul> |
| | descriptive | MHCVD | History of cerebrovascular disease<br>(e.g. TIA / Stroke) | nominal | ∘ Yes ∘ No |
| | descriptive | MHPVAD | Peripheral vascular/arterial disease | nominal | ∘ Yes ∘ No |
| | descriptive | MHASTH | Asthma or other chronic lung disease (except COPD) | nominal | ∘ Yes ∘ No |
| | descriptive | MHCOPD | Chronic obstructive pulmonary disease (COPD) | nominal | ∘ Yes ∘ No |
| | descriptive | MHSAP | Sleep apnoea | nominal | <ul><li>Yes ○ No</li></ul> |
| | descriptive | MHLIVR | Chronic liver disease | nominal | <ul><li>Yes ○ No</li></ul> |
| | descriptive | MHDIAM | Diabetes mellitus | nominal | <ul><li>Yes ○ No</li></ul> |
| | descriptive | MHANEM | Anemia | nominal | <ul><li>Yes ○ No</li></ul> |
| | descriptive | MHCNCR | Cancer | nominal | ∘ Yes ∘ No |
| | descriptive | MHHPLP | Hyperlipidemia | nominal | ∘ Yes ∘ No |
| | descriptive | МНСМВОТН | Other comorbidities | nominal | <ul><li>Yes ○ No</li></ul> |

| Data file,<br>identifier patient<br>display id full | | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|---|
| medical history | case case listing<br>for MHVHD = Yes | | Further specification of valvular heart disease (e.g. type, severity) | text | n.a. |
| | case listing<br>for MHCMBOTH<br>=Yes | СОСМВОТН | Specification of other comorbidities | text | n.a. |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



# 9.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

### 9.4. Exclusion of Particular Information

See general definitions in chapter 5.5.

No data are excluded from the specified analysis set and variables.

# 9.5. Descriptive Analyses

For specification "Notes = descriptive", see general definitions in chapter 5.1.

# 9.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 10. ADE and DD Endpoints - Implantation

### CIP chapter 7.2.2. Endpoints

In this study the number of adverse device effects and device deficiencies (DD) that occur in patients, users or other persons will be evaluated ...

- · Number of adverse device Effects / device deficiencies per number of implantations
- · Number of adverse device Effects / device deficiencies and per number of follow-up cases

ADEs will be adjudicated by an internal adjudication board, whereby the seriousness and device relatedness will be re-examined. If any amply documented external physical influence (e.g. accident, general power blackout) or medical AE caused the ADE, it does not contribute to this endpoint.

ADEs and device deficiencies are adjudicated by an internal adjudication board.

# 10.1. Analysis Set and Data Selection

All analyses are performed for patients in the implantation analysis set using a specific data selection before / at implantation  $^{15}$ .

#### 10.2. Variables

### Adjudicated Adverse Device Effects / Device Deficiencies

| Data file,<br>identifier<br>record id | Notes | Variable<br>name | Variable<br>label | Variable<br>Level | Nominal<br>values |
|---|---|---|---|---|---|
| internal adjudication | Case listing for AETYP | AETYP | Type of event | nominal | ∘ AE<br>∘ DD |
| | = AE | AESTDT | Onset date | date | n.a. |
| | | PRUCASE | Related use case | nominal | o Implementation<br>o PHD / Follow-up |
| | | DEIDV | Related investigational device | nominal | ∘ Renamic Neo programmer<br>∘ ECG cable PK-222-L |
| | | DIPRGSNR | Programmer serial number | text | n.a. |
| | | DIECBID | ESG cable ID | nominal | 01, 02,, 25 |
| | | AERELIDV | Adverse Event is related to the investigational device (device related ADE) | nominal | o Not related<br>o Unlikely<br>o Possible<br>o Probable<br>o Causal relationship |
| | | AESER | Adverse Event is serious | nominal | o Yes<br>o No |
| | | AERELSET | Adverse Event is relevant for<br>ADE/DD endpoint | nominal | ∘ Yes<br>∘ No |
| | | CORELSET | Please specify reson for No | text | n.a. |



 $<sup>^{15}</sup>$  analysis set imp SAR = Yes and PRUCASE = Implementation

| Data file,<br>identifier<br>record id | Notes | | Variable<br>label | Variable<br>Level | Nominal<br>values |
|---|---|---|---|---|---|
| internal<br>adjudication | Case listing<br>for AETYP | AETYP | Type of event | nominal | ∘ <b>AE</b><br>∘ DD |
| | = DD | DERCDT | Date of detection | date | n.a. |
| | | PRUCASE | Related use case | nominal | o Implementation<br>o PHD / Follow-up |
| | | DEIDV | Related investigational device | nominal | o Renamic Neo programmer<br>o ECG cable PK-222-L |
| | | DIPRGSNR | Programmer serial number | text | n.a. |
| | | DIECBID | ESG cable ID | nominal | 01, 02,, 25 |
| | | | Device dfficiency is relevant for ADE/DD endpoint | nominal | o Yes<br>o No |
| | | COADEDD | Please specify reson for No | text | n.a. |

| Data file,<br>identifier<br>patient display<br>id full | Notes | Variable<br>name | Variable<br>label | Variable<br>Level | Nominal<br>values |
|---|---|---|---|---|---|
| data SAR | descriprive | any ade SAR <sup>16</sup> | Any Adverse Device Effect<br>(serious or non-serious)<br>based on internal adjudication | nominal | o Yes<br>o No |
| data SAR | descriprive | any sade SAR <sup>17</sup> | Any Serious Adverse Device Effect based on internal adjudication | nominal | ∘ Yes<br>∘ No |
| data SAR | | any dd SAR <sup>18</sup> | Any Device Deficiency | nominal | ∘ Yes<br>∘ No |
| data SAR | descriprive | any ade dd SAR <sup>19</sup> | Any Adverse Device Effect<br>(serious or non-serious) or<br>Device Deficiency<br>based on internal adjudication | nominal | ∘ Yes<br>∘ No |
| data SAR | descriprive | n ade SAR <sup>20</sup> | Number of Adverse Device Effects<br>(serious or non-serious) based on internal<br>adjudication | metric to be reported as nominal | o1<br>o2<br> |
| data SAR | descriprive | n sade SAR <sup>21</sup> | Number of any Serious Adverse Device<br>Effects based on internal adjudication | metric to be reported as nominal | o1<br>o2<br> |
| data SAR | descriprive | n dd SAR <sup>22</sup> | Number of any Device Deficiencies based on internal adjudication | metric to be reported as nominal | o1<br>o2<br> |
| data SAR | descriprive | n ade dd SAR <sup>23</sup> | Number of any Adverse Device Effects<br>(serious or non-serious) and Device<br>Deficiencies based on internal adjudication | metric to be reported as nominal | o1<br>o2<br> |

```
16 If specific patient with AERELSET = Yes AND AESER = No
```

THEN any ade SAR = Yes ELSE any ade SAR = No

<sup>17</sup> If specific patient with AERELSET = Yes AND AESER = Yes

THEN any sade SAR = Yes ELSE any sade SAR = No

18 If specific patient with DEADEDD = Yes

THEN any dd SAR = Yes ELSE any dd SAR = No

19 If specific patient with AERELSET = Yes OR DEADEDD = Yes

THEN any ade dd AERELSET SAR = Yes

ELSE any ade dd SAR = No

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



<sup>&</sup>lt;sup>20</sup> Count number of events per patient with AERELSET = Yes AND AESER = No

<sup>&</sup>lt;sup>21</sup> Count number of events per patient with AERELSET = Yes AND AESER = Yes

<sup>&</sup>lt;sup>22</sup> Count number of events per patient with DEADEDD = Yes

<sup>&</sup>lt;sup>23</sup> Count number of events per patient with AERELSET = Yes OR DEADEDD = Yes

# 10.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

### 10.4. Exclusion of Particular Information

See general definitions in chapter 5.5. No data are excluded from the specified analysis set and variables.

# 10.5. Descriptive Analyses

For specification "Notes = descriptive", see general definitions in chapter 5.1.

# 10.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 11. ADE and DD Endpoints - PHD & follow-up

# CIP chapter 7.2.2. Endpoints

In this study the number of adverse device effects and device deficiencies (DD) that occur in patients, users or other persons will be evaluated ...

- · Number of adverse device Effects / device deficiencies per number of implantations
- · Number of adverse device Effects / device deficiencies and per number of follow-up cases

ADEs will be adjudicated by an internal adjudication board, whereby the seriousness and device relatedness will be re-examined. If any amply documented external physical influence (e.g. accident, general power blackout) or medical AE caused the ADE, it does not contribute to this endpoint.

ADEs and device deficiencies are adjudicated by an internal adjudication board.

### 11.1. Analysis Set and Data Selection

All analyses are performed for patients in the PHD & follow-up analysis set using a specific data selection after implantation<sup>24</sup>.

All analyses from chapter 10 ADE and DD Endpoints - Implantation are repeated for these data.

<sup>&</sup>lt;sup>24</sup> analysis set PHD FUP SAR = Yes and PRUCASE = PHD / Follow-up



# 12. Implantation & PSA

# CIP chapter 7.5 Further data of interest

During implantation and follow-ups additional data on safety, performance and usability of the Renamic Neo system and accessories will be collected.

· Use and assessment of PSA functionality (sensing, pacing and impedance tests)...

# 12.1. Analysis Set

All analyses are performed for patients in the implantation analysis set<sup>25</sup>.

#### 12.2. Variables

### <u>Used Programmer Features: Pacing System Analyzer (PSA)</u>

| Data file | Notes | \/a wia la la | Variable | Maniah I- | Neminal |
|---|---|---|---|---|---|
| Data file, | Notes | Variable | Variable | | Nominal |
| identifier patient | | name | label | Level | values |
| display id full | 1 | DD 114DC 4 | W | | |
| implantation psa | descriptive | PRIMPSA | Was the PSA functionality used | nominal | |
| | | | during implantation | | o No |
| | descriptive with | QSPLRAS | Polarity selection and | nominal | oused successfully |
| | "not used" | | documentation | | oused, but not successfully |
| | handled as missing | | | | o not used |
| | descriptive# | QSPLRSPR | NEW: Polarity: | nominal | <ul><li>Yes, with Adverse Event</li></ul> |
| | | | Did you notice any problem | | <ul><li>Yes, without Adverse Event</li></ul> |
| | | | | | o No problem detected |
| | descriptive with | QSSAAS | Sensing amplitude | nominal | o used successfully |
| | "not used" | | | | oused, but not successfully |
| | handled as missing | | | | o not used |
| | descriptive# | QSSAPRB | NEW: Sensing amplitude: Did | nominal | <ul><li>Yes, with Adverse Event</li></ul> |
| | | | you notice any problem | | o Yes, without Adverse Event |
| | | | | | o No problem detected |
| | descriptive with | QSPTAS | Pacing threshold | nominal | o used successfully |
| | "not used" | _ | | | oused, but not successfully |
| | handled as missing | | | | o not used |
| | descriptive# | QSPRPRB | NEW: Pacing threshold: | nominal | o Yes, with Adverse Event |
| | | | Did you notice any problem | | o Yes, without Adverse Event |
| | | | , , , | | o No problem detected |
| | descriptive with | QSPITAS | Impedance test | nominal | o used successfully |
| | "not used" | | | | oused, but not successfully |
| | handled as missing | | | | o not used |
| | descriptive# | | NEW: Impedance test: | nominal | o Yes, with Adverse Event |
| | | | Did you notice any problem | | o Yes, without Adverse Event |
| | | | | | o No problem detected |
| | descriptive with | QSPNSAS | Phrenic Nerve Stimulation (PNS) | nominal | oused successfully |
| | "not used" | Qu'illorie | test and documentation | | oused, but not successfully |
| | handled as missing | | | | o not used |
| | descriptive# | | NEW: PNS test: | nominal | o Yes, with Adverse Event |
| | accorpance | QUI NOI NO | Did you notice any problem | | o Yes, without Adverse Event |
| | | | 2.5 , 55 Hotioc arry problem | | No problem detected |
| | descriptive with | QSBSAS | Burst stimulation | nominal | o used successfully |
| | "not used" | QUUUNU | if performed in routine care | | oused, but not successfully |
| | handled as missing | | performed in roudine care | | o not used |
| | descriptive# | QSBSPRB | NEW: Burst stimulation: | nominal | o Yes, with Adverse Event |
| | uescriptive# | QSBSFKB | Did you notice any problem | Hominal | o Yes, without Adverse Event |
| | | | Did you notice any problem | | o No problem detected |
| | | | | | ono problem detected |

# If preceding variable = "used successfully" then impute missing data with "used successfully".

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



 $<sup>^{25}</sup>$  analysis set imp SAR = Yes

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier patient | Notes | name | label | Level | values |
| display id full | | Tidiric . | | 20101 | Values |
| implantation psa | case listing for QSPLRAS = used, but not successfully OR QSPLRSPR = Yes, with Adverse Event OR QSPLRSPR = Yes, without Adverse Event including programmer serial number DIPRGSNR (see chapter15.1) | | NEW: Polarity amplitude:<br>Please specify reason for<br>unsuccessful use | text | |
| | case listing for QSSAAS = used, but not successfully OR QSSAPRB = Yes, with Adverse Event OR QSSAPRB = Yes, without Adverse Event including programmer serial number DIPRGSNR (see chapter15.1) | COSAAS | NEW: Sensing amplitude:<br>Please specify reason for<br>unsuccessful use | text | |
| | case listing for QSPTAS = used, but not successfully OR QSPRPRB = Yes, with Adverse Event OR QSPRPRB = Yes, without Adverse Event including programmer serial number DIPRGSNR (see chapter15.1) | COPTAS | NEW: Pacing threshold:<br>Please specify reason for<br>unsuccessful use | text | |
| | case listing for QSPITAS = used, but not successfully OR QSPITPRB = Yes, with Adverse Event OR QSPITPRB = Yes, without Adverse Event including programmer serial number DIPRGSNR (see chapter15.1) | COPITAS | NEW: Impedance test:<br>Please specify reason for<br>unsuccessful use | text | |
| | case listing for QSPNSAS = used, but not successfully OR QSPNSPRB = Yes, with Adverse Event OR QSPNSPRB = Yes, without Adverse Event including programmer serial number DIPRGSNR (see chapter15.1) | COPNSAS | NEW: PNS test: Please<br>specify reason for<br>unsuccessful use | text | |
| | case listing for QSBSAS= used, but not successfully OR QSBSPRB = Yes, with Adverse Event OR QSBSPRB = Yes, without Adverse Event including programmer serial number DIPRGSNR (see chapter15.1) | COBSAS | NEW: Burst stimulation:<br>Please specify reason for<br>unsuccessful use | text | |

# Used Measurement Mode: Pacing System Analyzer (PSA)

| Data file,<br>identifier patient<br>display id full | Notes | | | | Nominal<br>values |
|---|---|---|---|---|---|
| mprantación pod | | | dual and triple chamber devices are measured consecutively in single-chamber mode, e.g. VVI) | nominal | o Yes<br>o No |
| | descriptive | DUDCHM | Dual chamber mode (e.g. VDD RV) | nominal | o Yes<br>o No |
| | descriptive | DUTCHM | Triple chamber mode (e.g. DDI BiV) | nominal | ∘Yes<br>∘No |
| | descriptive | | Was radio frequency (RF) electrosurgical equipment used while the PSA was connected to the pacing lead(s) | nominal | o Yes<br>o No |

| Data file,<br>identifier patient<br>display id full | | | Variable<br>Level | Nominal<br>values |
|---|---|---|---|---|
| implantation psa | case listing for DURFSE = Yes | Please specify type of RF surgical equipment used | text | |



# 12.1. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 12.2. Exclusion of Particular Information

See general definitions in chapter 5.5.

No data are excluded from the specified analysis set and variables.

# 12.3. Descriptive Analyses

For specification "Notes = descriptive", see general definitions in chapter 5.1.

# 12.4. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 13. General Assessments - Implantation

### CIP chapter 7.5 Further data of interest

During implantation and follow-ups additional data on safety, performance and usability of the Renamic Neo system and accessories will be collected.

- · Use and assessment of PSA functionality (sensing, pacing and impedance tests)
- · Success of adequate programming of the implant
- · Evaluation of interrogation of the implant including RF telemetry
- · Overall assessment of device hardware or software performance including battery use
- Data export evaluation (used connectivity, destination, printing)

# 13.1. Analysis Set and Data Selection

All analyses are performed for patients in the implantation analysis set using a specific data selection before / at implantation<sup>26</sup>.

| Data file, identifier | Notes | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|---|
| patient display | | name | label | level | |
| id full & | | | | | |
| autom SVTYP | | | | | |
| general | No report | autom SVTYP | Visit type | nominal | o Implantation |
| assessments | | | | | o Pre-hospital discharge follow-up (PHD) |
| | | | | | o Regular follow-up after PHD |

 $<sup>^{26}</sup>$  analysis set imp SAR = Yes Data selection for general assessments with autom SVTYP = implantation



# Used Programmer Features: Implant

| Data file, identifier | Notes | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|---|
| patient display | | name | label | level | |
| id full & autom SVTYP | | | | | |
| general | descriptive | QSPGHAS | Programmer head (PGH) | nominal | o used successfully |
| assessments | | | telemetry | | oused, but not successfully |
| (see Analysis Set<br>and Data Selection) | descriptive# | | Did you notice any problem*<br>(see definition above) with<br>usage of programmer head<br>telemetry | | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |
| | descriptive<br>with "not used" and<br>"not available"<br>handled as missing | QSRFTAS | RF telemetry for implant interrogation | nominal | o used successfully o used, but not successfully o not used o not available for implant by default |
| | descriptive# | QSRFTPRB | Did you notice any problem*<br>(see definition above) with<br>usage of RF telemetry for<br>implant interrogation | | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |
| | descriptive with<br>"not used"<br>handled as missing | QSSAAS | Sensing amplitude | nominal | o used successfully<br>o used, but not successfully<br>o not used |
| | descriptive# | QSSAPRB | (see definition above) with usage of sensing amplitude | | <ul><li>Yes, with Adverse Event</li><li>Yes, without Adverse Event</li><li>No problem detected</li></ul> |
| | descriptive<br>with "not used"<br>handled as missing | QSPTAS | Pacing threshold | nominal | o used successfully<br>o used, but not successfully<br>o not used |
| | descriptive# | QSPRPRB | Did you notice any problem*<br>(see definition above) with<br>usage of pacing threshold | | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |
| | descriptive<br>with "not used"<br>handled as missing | QSPITAS | Impedance test | | o used successfully o used, but not successfully o not used |
| | descriptive# | QSPITPRB | Did you notice any problem*<br>(see definition above) with<br>usage of impedance test | nominal | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |
| | descriptive<br>with "not used" OR<br>VectorOpt not<br>available"<br>handled as missing | QSDFPAS | LV Pacing threshold and PNS measurement for different polarities | nominal | o used successfully o used, but not successfully o not used o VectorOpt not available for CRT implant |
| | descriptive# | | Did you notice any problem*<br>(see definition above) with<br>usage of LV Vector Opt<br>function | | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |
| | descriptive<br>with "not done"<br>handled as missing | QSPRGAS | Programming of the implant | nominal | o device successfully<br>programmed<br>o device not successfully<br>programmed<br>o not done |
| | descriptive# | | Did you notice any problem*<br>(see definition above) with<br>usage of programming<br>of the implant function | | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |
| | descriptive<br>with "not used"<br>handled as missing | QSDFTAS | DFT (Defibrillation Threshold<br>Testing) if performed in<br>routine care | nominal | o used successfully o used, but not successfully o not used |
| | descriptive# | QSDFTPRB | | nominal | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |

# If preceding variable = "used successfully" or "device successfully programmed" then impute missing data with "Used successfully".

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



| Data file, identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient display | | name | label | level | values |
| id full & | | | | | |
| autom SVTYP | | | | | |
| general | case listing for | COPGHAS | Please specify reason for | text | |
| assessments | QSPGHAS = used, but not successfully OR | | unsuccessful use of | | |
| (see Analysis Set | QSPGHPRB = Yes, with Adverse Event OR | | programmer head telemetry | | |
| and Data Selection) | QSPGHPRB = Yes, without Adverse Event | | | | |
| | including programmer serial number | | | | |
| | DIPRGSNR (see chapter15.1) | | - Is | | |
| | case listing for | CORFTAS | Please specify reason | text | |
| | QSRFTAS = used, but not successfully OR | | for unsuccessful use of RF telemetry | | |
| | QSRFTPRB = Yes, with Adverse Event OR<br>QSRFTPRB = Yes, without Adverse Event | | for implant interrogation | | |
| | including programmer serial number | | I implant interrogation | | |
| | DIPRGSNR (see chapter15.1) | | | | |
| | case listing for | COSAAS | Please specify reason | text | |
| | QSSAAS = used, but not successfully OR | COSAAS | for unsuccessful use | CCAC | |
| | QSSAPRB = Yes, with Adverse Event | | of sensing amplitude | | |
| | QSSAPRB = Yes, without Adverse Event | | | | |
| | including programmer serial number | | | | |
| | DIPRGSNR (see chapter15.1) | | | | |
| | case listing for | COPTAS | Please specify reason | text | |
| | QSPTAS = used, but not successfully OR | | for unsuccessful use | | |
| | QSPRPRB = Yes, with Adverse Event OR | | of pacing threshold | | |
| | QSPRPRB = Yes, without Adverse Event | | | | |
| | including programmer serial number DIPRGSNR (see chapter15.1) | | | | |
| | case listing for | COPITAS | Please specify reason | text | |
| | QSPITAS = used, but not successfully OR | 601117.5 | for unsuccessful use | COAC | |
| | QSPITPRB = Yes, with Adverse Event OR | | of impedance test | | |
| | QSPITPRB = Yes, without Adverse Event | | | | |
| | including programmer serial number | | | | |
| | DIPRGSNR (see chapter15.1) | | | | |
| | case listing for | CODFPAS | Please specify reason | text | |
| | QSDFPAS = used, but not successfully OR | | for unsuccessful use | | |
| | QSDFPPRB = Yes, with Adverse Event OR | | of LV Vector Opt function | | |
| | QSDFPPRB = Yes, without Adverse Event | | | | |
| | including programmer serial number | | | | |
| | DIPRGSNR (see chapter15.1) | CODDCAC | Diana anadifu maaan | tout | |
| | case listing for<br>QSPRGAS = used, but not successfully OR | COPRGAS | Please specify reason for unsuccessful | text | |
| | QSPRGPRB = Yes, with Adverse Event OR | | programming | | |
| | QSPRGPRB = Yes, without Adverse Event | | of the implant | | |
| | including programmer serial number | | | | |
| | DIPRGSNR (see chapter15.1) | | | | |
| | case listing for | CODFTAS | Please specify reason | text | |
| | QSDFTAS = used, but not successfully OR | | for unsuccessful use | | |
| | QSDFTPRB = Yes, with Adverse Event OR | | of DFT | | |
| | QSDFTPRB = Yes, without Adverse Event | | | | |
| | including programmer serial number | | | | |
| | DIPRGSNR (see chapter15.1) | | | | |



# **Accuracy of PSA Measurements**

The analyses specified in this sub-chapter have to be performed for the implantation analysis set only.

| Data file, identifier patient display id full & autom SVTYP | Notes | <br>Variable<br>label | Variable<br>Ievel | Nominal values |
|---|---|---|---|---|
| general<br>assessments<br>(see Analysis Set and<br>Data Selection) | descriptive with<br>"no comparison<br>possible"<br>handled as missing | Are PSA measurement results (sensitivity, pacing threshold, impedance) sufficiently accurate, compared to the measurement results of the implanted device | | o Yes<br>o No<br>o no comparison possible |

| Data file, identifier patient display id full & autom SVTYP | Notes | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|
| assessments<br>(see Analysis Set and<br>Data Selection) | case listing for DUPSAAS = No OR DUPSAAS = no comparison possible including programmer serial number DIPRGSNR (see chapter15.1) | Please specify<br>No / no comparison<br>possible | text | |



# Used Programmer Features: Data export

| Data file, identifier patient display id full & autom SVTYP | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| general<br>assessments | descriptive | PRDEXP | Was data export performed | nominal | ∘ Yes<br>∘ No |
| (see Analysis Set and Data Selection) | | DULAN01 | NEW: Connectivity: LAN | nominal | o Yes<br>o No |
| , | | DUWLAN01 | NEW: Connectivity: WLAN | nominal | o Yes<br>o No |
| | | DUUSB01 | NEW: Connectivity: USB | nominal | o Yes<br>o No |
| | | QSCNNAS | Was connectivity used successfully | nominal | ∘ Yes<br>∘ No |
| | | QSCNNPRB<br># | <b>NEW: Connectivity:</b> Did you notice any problem* (see definition above) | nominal | o Yes<br>o No problem detected |
| | | DUNTSH | <b>NEW: Data export:</b> Network share (for EHR) | nominal | o Yes<br>o No |
| | | DUUSBS | NEW: Data export: USB stick | nominal | ∘Yes<br>∘No |
| | | DUOTH | NEW: Data export: Other | nominal | ∘ Yes<br>∘ No |
| | | PRDEXPAS | Was data export successful | nominal | ∘Yes<br>∘No |
| # T6 dia | | # | <b>NEW: Data export:</b> Did you notice any problem* (see definition above) | | o Yes<br>o No problem detected |

<sup>#</sup> If preceding variable = "Yes" then impute missing data with "Used successfully".

| Data file, identifier patient display id full & autom SVTYP | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| general<br>assessments<br>(see Analysis Set<br>and Data Selection) | case listing for<br>QSCNNAS = No OR<br>QSCNNPRB = Yes | | <b>NEW: Connectivity:</b> Please specify reason for unsuccessful use | text | |
| | case listing for<br>PRDEXPAS = No OR<br>QSDEXPPR = Yes | | <b>NEW: Data export:</b> Please specify reason for unsuccessful use | text | |
| | case listing for<br>DUOTH = Yes | СООТН | <b>NEW: Data export:</b> Please specify Other | text | |



# **Used Programmer Features: Printing**

| Data file, identifier<br>patient display<br>id full &<br>autom SVTYP | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| general<br>assessments | decriptive | PRPRNT | Was printing performed | nominal | ∘ Yes<br>∘ No |
| (see Analysis Set and Data Selection) | | DULAN02 | NEW: Printing LAN | nominal | o Yes<br>o No |
| | | DUWLAN02 | NEW: Printing WLAN | nominal | o Yes<br>o No |
| | | DUUSB02 | NEW: Printing USB | nominal | o Yes<br>o No |
| | | QSPRNTAS | Was printing successful | | ∘Yes<br>∘No |
| | QSPRN<br># | • | <b>NEW: Printing:</b> Did you notice any problem* (see definition above) | nominal | o Yes<br>o No problem detected |
| | | DUPRNTTY | Please specify which printer type was used | nominal | |

<sup>#</sup> If preceding variable = "Yes" then impute missing data with "Used successfully".

| Data file, identifier | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| patient display | | name | label | level | values |
| id full & | | | | | |
| autom SVTYP | | | | | |
| general | case listing for | CODEXPAS | NEW: Printing: Please specify reason for | text | |
| assessments | QSPRNTAS = No OR | | unsuccessful use | | |
| (see Analysis Set | QSPRNTPR = Yes | | | | |
| and Data Selection) | - | | | | |

### **Used Programmer Features: Battery**

| Data file, identifier patient display id full & autom SVTYP | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| general<br>assessments<br>(see Analysis Set<br>and Data Selection) | descriptive with "not used" handled as missing | PRPRGB | Was the programmer used with the battery as power supply (without power cable, usage is optional) | | o used successfully<br>o used, but not successfully<br>o not used |
| | descriptive,<br>if PRPRGB = "successfully used"<br>then impute missing QSPRGBPR<br>with "No problem detected".# | QSPRGBPR | NEW: battery:<br>Did you notice<br>any problem*<br>(see definition<br>above) | nominal | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |

# # If preceding variable = "Used successfullyes" then impute missing data with "Used successfully".

| Data file, identifier patient display | Notes | | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| id full & | | name . | label . | 10.00 | values |
| autom SVTYP | | | | | |
| (see Analysis Set and Data Selection) | case listing for PRPRGB= used, but not successfully OR QSPRGBPR = Yes, with Adverse Event OR QSPRGBPR = Yes, without Adverse Event including programmer serial number DIPRGSNR (see chapter15.1) | | NEW: Battery: Please<br>specify reason for<br>unsuccessful use | text | |





# Assessment of Programmer Features

| Data file,<br>identifier<br>patient display<br>id full &<br>autom SVTYP | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| general assessments (see Analysis Set and Data Selection) | | QSCNSAS | Are the connectivity settings<br>(e.g. WLAN, LAN, printer)<br>easy / difficult to find | nominal | o Very easy o Easy o Adequate o Somewhat difficult o Very difficult |
| | | QSPSAPAS | Are the PSA parameters<br>(e.g. amplitude, basic rate, mode)<br>easy / difficult to find | nominal | o Very easy o Easy o Adequate o Somewhat difficult o Very difficult |
| | | QSPGPV | Is the range of programmable variables for connectivity settings (e.g. WLAN, LAN, printer) sufficient | nominal | o Yes<br>o No |
| | | QSRGPSA | Is the range of the PSA parameters<br>(e.g. amplitude, basic rate, mode)<br>sufficient for the treatment of the patient | nominal | oYes<br>oNo |
| | | (Note:<br>No missing | Did you notice any problems* (including IEGM and ECG recording) which are not mentioned yet relating to the device hardware or software | nominal | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |

| Data file, identifier patient display id full & autom SVTYP | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| general<br>assessments<br>(see Analysis Set<br>and Data Selection) | case listing for QSCNSAS = Somewhat difficult OR QSCNSAS = Very difficult including programmer serial number DIPRGSNR (see chapter15.1) | COCNSAS | NEW: Data export:<br>Please specify<br>Somewhat difficult /<br>Very difficult | text | |
| | case listing for QSPSAPAS = Somewhat difficult OR QSPSAPAS = Very difficult including programmer serial number DIPRGSNR (see chapter15.1) | COPSAPAS | NEW: Printing:<br>Please specify<br>Somewhat difficult /<br>Very difficult | text | |
| | case listing for QSPGPV = No<br>including programmer serial number<br>DIPRGSNR (see chapter15.1) | COPGPV | NEW: Battery:<br>Please specify in case of NO | text | ••• |
| | case listing for QSRGPSA = No including programmer serial number DIPRGSNR (see chapter15.1) | CORGPSA | Please specify in case of NO | text | |
| | Case listing for all non-missing data<br>including programmer serial number<br>DIPRGSNR (see chapter15.1) | general<br>comment | General comment | text | |

| Data file, identifier patient display id full | 1,1000 | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| data SAR | case listing for any reported problem: QSPGHPRB, QSRFTPRB, QSSAPRB, QSPRPRB, QSPITPRB, QSDFPPRB, QSPRGPRB, QSDFTPRB contain "Yes"; DUPSAAS = No, QSCNNPRB, QSDEXPPR, QSPRNTPR, QSPRGBPR QSANYPRB contain "Yes" | | Program<br>mer<br>serial<br>number | text | |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.


## 13.1. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 13.2. Exclusion of Particular Information

See general definitions in chapter 5.5.

No data are excluded from the specified analysis set and variables.

# 13.3. Descriptive Analyses

For specification "Notes = descriptive", see general definitions in chapter 5.1.

### 13.4. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 14. General Assessments - PHD & Follow-up

#### CIP chapter 7.5 Further data of interest

During implantation and follow-ups additional data on safety, performance and usability of the Renamic Neo system and accessories will be collected.

- · Use and assessment of PSA functionality (sensing, pacing and impedance tests)
- · Success of adequate programming of the implant
- · Evaluation of interrogation of the implant including RF telemetry
- · Overall assessment of device hardware or software performance including battery use
- · Data export evaluation (used connectivity, destination, printing)

### 14.1. Analysis Set and Data Selection

All analyses are performed for patients in the PHD and follow-up analysis set using a specific data selection after implantation<sup>27</sup>.

All analyses from chapter 13 Devices and Accessories - Implantation are repeated for these data. However, "implantation" will be replaced by "PHD & follow-up".

<sup>&</sup>lt;sup>27</sup> analysis set PHD FUP SAR = Yes
Data selection for general assessments with autom SVTYP ≠ implantation



# 15. Devices and Accessories - Implantation

### CIP chapter 7.5 Further data of interest

General information

- · Implant type and model, all other implanted devices
- · Lead model and programmer software version

During implantation and follow-ups additional data on safety, performance and usability of the Renamic Neo system and accessories will be collected.

... Information on additionally used accessories or other implanted cardiac devices

### 15.1. Analysis Set and Data Selection

All analyses are performed for patients in the implantation analysis set using a specific data selection before / at implantation<sup>28</sup>.

#### **Implanted Devices**

| Data file, identifier patient display id full & DIDVTYP | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| device log details | No report | DIDVTYP | General type of<br>device/lead | | o Pacemaker (single/dual chamber) o ICD (single/dual chamber) o CRT-P device o CRT-D device o ICM (Insertable Cardiac Monitor) o RA lead o RV lead o LV lead o VCS lead |
| | | DTDVSTAT | Status of device | | o Implanted and active o Deactivated but still implanted o Explanted and returned to manufacturer o Explanted and discarded o Attempted implantation, then returned o Attempted implantation, then discarded |
| | | DIDVMDL | Device / lead model | text | <b></b> |

| Data file, identifier patient display id full | | | | | Nominal values |
|---|---|---|---|---|---|
| data SAR | descriptive | device model SAR <sup>29</sup> | Device model | text | |

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.

= DIDVMDL

device model SAR



<sup>&</sup>lt;sup>28</sup> analysis set imp SAR = Yes
Data selection for accessory log details with SVTYP = implantation

| Data file, identifier patient display id full | | | | | Nominal values |
|---|---|---|---|---|---|
| data SAR | descriptive | lead RA model SAR <sup>30</sup> | RA lead model | text | |
| | | 24 | RV lead model | text | |
| | | lead LV model SAR32 | LV lead model | text | |
| | | lead VSC model SAR33 | VCS lead model | text | |

#### Renamic Neo and software

| Data file, identifier patient display id full & autom SVTYP | | Variable<br>name | | Variable<br>Ievel | Nominal values |
|---|---|---|---|---|---|
| accessory log details | No report | SVTYP | Visit type | | o Implantation<br>o Pre-hospital discharge<br>o Follow-up |

| Data file, identifier<br>patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | Notes | | | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| accessory log details | Selection DIPRGMDL = | DIPRGSNR | Programmer serial number | text | |
| | Renamic Neo;<br>no report | DISFTVER | Programmer software version | | NEO 2004.A |

Note: In case of any reported problem, the serial number DIPRGSNR of the Renamic Neo, which was used for the specific investigation for a specific patient (or programmers in case more than one programmer were used), will be reported together with the patient id patient display id full.

| Data file, identifier<br>DIPRGSNR | Variable<br>name | | | Nominal<br>values |
|---|---|---|---|---|
| renamicneo SAR | renamicneo SAR <sup>34</sup> | performed with specific Renamic | metric to be reported as nominal | 1 2 |

| / | | Variable | | | Nominal |
|---|---|---|---|---|---|
| identifier patient | | name | label | Level | values |
| display id full | | | | | |
| data SAR | descriptive | n renamicneo imp SAR <sup>35</sup> | Number of Renamic Neo | metric to be | 1 |
| | | | programmers used during | reported as | 2 |
| | | | implantation | nominal | |
| | | n renamicneo imp | Number of Renamic Neo | metric to be | 1 |
| | | NEO2004A SAR <sup>36</sup> | programmers with software NEO | reported as | 2 |
| | | | 2004.A used during implantation | nominal | |

Patient-specific data for lead RA model SAR = DIDVTYP = RA lead AND DTDVSTAT = Implanted and active DIDVMDL

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



Patient-specific data for lead RV model SAR = DIDVTYP = RV lead AND DTDVSTAT = Implanted and active DIDVMDL

Patient-specific data for lead LV model SAR = DIDVTYP = LV lead AND DTDVSTAT = Implanted and active DIDVMDL

Patient-specific data for lead VCS model SAR = DIDVTYP = VCS lead AND DTDVSTAT = Implanted and active DIDVMDL

<sup>&</sup>lt;sup>34</sup> Count different patient display id full per DIPRGSNR from accessory log details with SVTYP = Implantation

<sup>35</sup> Count different DIPRGSNR per patient display id full for SVTYP = Implantation

 $<sup>^{36}</sup>$  Count different DIPRGSNR with DISFTVER = "NEO 2004.A" per patient display id full for SVTYP = Implantation

#### ECG cable

| Data file, identifier | Notes | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|---|
| patient display id full & | | name | label | level | |
| SVTYP & | | | | | |
| helpvar model & | | | | | |
| DIPRGSNR | | | | | |
| accessory log details | no report | DIECBMDL | ECG cable model | nominal | o PK-222-L ECG cable |
| (see Analysis Set and | | | | | o PK-222 EU / 2.8 m ECG cable |
| Data Selection) | | QSECBAS | Usage of ECG cable | nominal | o used successfully |
| | | | | | oused, but not successfully |
| | | QSECBPRB | Did you notice any | nominal | o Yes, with Adverse Event |
| | | | problems related to | | <ul><li>Yes, without Adverse Event</li></ul> |
| | | | ECG cable | | <ul> <li>No problem detected</li> </ul> |

| Data file, identifier<br>patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | Notes | <br>Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|
| (see Analysis Set and Data Selection) | case listing for QSECBAS = used, but not successfully OR QSECBPRB = Yes, with Adverse Event OR QSECBPRB = Yes, without Adverse Event including programmer serial number DIPRGSNR (see note before) | NEW: ECG cable at investigattion: Please specify reason for unsuccessful use | text | |

| Data file,<br>identifier patient<br>display id full | Notes | Variable<br>name | Variable<br>label | Variable<br>Level | Nominal values |
|---|---|---|---|---|---|
| | | n ecgcable PK<br>imp SAR <sup>37</sup> | Number of PK<br>ECG cables used during<br>implantation | metric to be<br>reported as<br>nominal | o 1<br>o 2<br> |
| | | n ecgcable PK222L<br>imp SAR <sup>38</sup> | Number of PK-222-L<br>ECG cables used during<br>implantation | metric to be<br>reported as<br>nominal | o 1<br>o 2<br>o |
| | | n ecgcable PK222EU<br>imp SAR <sup>39</sup> | Number of PK-222-EU<br>ECG cables used during<br>implantation | metric to be reported as nominal | o 1<br>o 2<br> |
| | | n ecgcable nosucccess<br>imp SAR <sup>40</sup> | Number of ECG cables<br>not successfully used during<br>implantation | metric to be<br>reported as<br>nominal | o1<br>o2 |
| | | n ecgcable problem<br>imp SAR <sup>41</sup> | Number of ECG cables with any<br>problem used during<br>implantation | metric to be<br>reported as<br>nominal | o 1<br>o 2 |

<sup>&</sup>lt;sup>41</sup> Count QSECBPRB = "Yes, with Adverse Event" OR "Yes, without Adverse Event" per patient display id full



 $<sup>^{37}</sup>$  Count DIECBMDL = "PK-222-L ECG cable" OR "PK-222 EU / 2.8 m ECG cable" per patient display id full

<sup>38</sup> Count DIECBMDL = "PK-222-L ECG cable" per patient display id full

<sup>&</sup>lt;sup>39</sup> Count DIECBMDL = "PK-222 EU / 2.8 m ECG cable" per patient display id full

 $<sup>^{40}</sup>$  Count QSECBAS = "used, but not successfully" per patient display id full

### Electrode clip

| Data file, identifier | Notes | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|---|
| patient display id full & SVTYP & | | name | label | level | |
| helpvar model & DIPRGSNR | | | | | |
| accessory log details | no report | DIELDCMD | Electrode clip model | nominal | o PK Electrode Clip |
| (see Analysis Set and Data Selection) | | QSELDCAS | Usage of electrode clip | I . | o used successfully o used, but not successfully |
| | | QSELDCPR | Did you notice any problems related to electrode clip | | <ul><li>Yes, with Adverse Event</li><li>Yes, without Adverse Event</li><li>No problem detected</li></ul> |

| Data file, identifier | Notes | | | | Nominal |
|---|---|---|---|---|---|
| patient display id full & SVTYP & | | name | label | level | values |
| helpvar model & DIPRGSNR | | | | | |
| Data Selection) | case listing for QSELDCAS = used, but not successfully OR QSELDCPR = Yes, with Adverse Event OR QSELDCPR = Yes, without Adverse Event including programmer serial number DIPRGSNR (see note before) | | NEW: Electrode<br>clip: Please specify<br>reason for<br>unsuccessful use | text | |

| | | Variable | | | Nominal |
|---|---|---|---|---|---|
| identifier patient<br>display id full | | name | label | Level | values |
| data SAR | descriptive | | | metric to be | 01 |
| | | | 3 | reported as<br>nominal | o <b>2</b><br> |
| | | n elclip pk nosucccess imp SAR43 | | metric to be | o <b>1</b> |
| | | | , | reported as | o <b>2</b> |
| | | | implantation | nominal | |
| | | n elclip pk problem imp SAR44 | Number of used PK electrode | metric to be | 01 |
| | | | clips with any problem during | reported as | o <b>2</b> |
| | | | implantation | nominal | |

<sup>44</sup> Count QSELDCPR = "Yes, with Adverse Event" OR "Yes, without Adverse Event" per patient display id full



<sup>&</sup>lt;sup>42</sup> Count DIELDCMD = "PK Electrode Clip" per patient display id full

<sup>&</sup>lt;sup>43</sup> Count QSELDCAS = "used, but not successfully" per patient display id full

### Patient cable

| Data file, identifier<br>patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | Notes | Variable<br>name | | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| accessory log details<br>(see Analysis Set and<br>Data Selection) | no report | DIPCBMDL | Patient cable model | | o Patient cable PK-141 o Patient cable PK-67-S o Patient cable PK-67-L o Patient cable PK-155 |
| | | QSPCBAS | Usage of patient cable | nominal | oused successfully<br>oused, but not successfully |
| | | QSPCBPRB | Did you notice any<br>problems related to<br>patient cable | nominal | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |

| Data file, identifier<br>patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | | | | Nominal<br>values |
|---|---|---|---|---|
| , 3 | case listing for QSPCBAS = used, but not successfully OR QSPCBPRB = Yes, with Adverse Event OR QSPCBPRB = Yes, without Adverse Event including programmer serial number DIPRGSNR (see note before) | NEW: Patent<br>cable: Please<br>specify reason for<br>unsuccessful use | text | |



| Data file,<br>identifier patient<br>display id full | Variable<br>name | Variable<br>label | Variable<br>Level | Nominal<br>values |
|---|---|---|---|---|
| data SAR | n patcable PK imp SAR <sup>45</sup> | Number of patient cables<br>PK used during implantation | metric to be<br>reported as<br>nominal | o 1<br>o 2<br> |
| | n patcable PK141 imp SAR <sup>46</sup> | Number of patient cables<br>PK-141 used during<br>implantation | metric to be reported as nominal | o 1<br>o 2<br>o |
| | n patcable PK67S imp SAR <sup>47</sup> | Number of patient cables<br>PK-67-S used during<br>implantation | metric to be<br>reported as<br>nominal | o1<br>o2<br> |
| | n patcable PK67L imp SAR <sup>48</sup> | Number of patient cables<br>PK-67-L used during<br>implantation | metric to be reported as nominal | o1<br>o2<br> |
| | n patcable PK155 imp SAR <sup>49</sup> | Number of patient cables<br>PK-155 used during<br>implantation | metric to be<br>reported as<br>nominal | o 1<br>o 2<br> |
| | n patcable nosuccess imp SAR <sup>50</sup> | | metric to be<br>reported as<br>nominal | ∘1<br>∘2<br> |
| | n patcable problem imp SAR <sup>51</sup> | Number of used patient cables with any problem during implantation | metric to be<br>reported as<br>nominal | ∘1<br>∘2<br> |

BIOTRONIK excellence for life

<sup>&</sup>lt;sup>45</sup> Count DIPCBMDL = "Patient cable PK-141" OR "67-S" OR "67-L" OR "155" per patient display id full

<sup>&</sup>lt;sup>46</sup> Count DIPCBMDL = "Patient cable PK-141" per patient display id full

 $<sup>^{47}</sup>$  Count DIPCBMDL = "Patient cable PK-67-S" per patient display id full

<sup>&</sup>lt;sup>48</sup> Count DIPCBMDL = "Patient cable PK-67-L" per patient display id full

<sup>&</sup>lt;sup>49</sup> Count DIPCBMDL = "Patient cable PK-155" per patient display id full

<sup>&</sup>lt;sup>50</sup> Count QSPCBAS = "used, but not successfully" per patient display id full

<sup>&</sup>lt;sup>51</sup> Count QSPCBPRB = "Yes, with Adverse Event" OR "Yes, without Adverse Event" per patient display id full

#### Patient adapter

| Data file, identifier<br>patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | Notes | | | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| accessory log details<br>(see Analysis Set and<br>Data Selection) | no report | DIPADMDL | Patient adapter model | nominal | o Patient adapter PA-1-B<br>o Patient adapter PA-1-C<br>o Patient adapter PA-2 |
| | | • | Usage of patient adapter | nominal | o used successfully o used, but not successfully |
| | | | Did you notice any problems related to patient adapter | nominal | o Yes, with Adverse Event<br>o Yes, without Adverse Event<br>o No problem detected |

| Data file, identifier<br>patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | Notes | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|
| accessory log details<br>(see Analysis Set and<br>Data Selection) | case listing for QSPADAS = used, but not successfully OR QSPADPRB = Yes, with Adverse Event OR QSPADPRB = Yes, without Adverse Event including programmer serial number DIPRGSNR (see note before) | NEW: Patent<br>adapter: Please<br>specify reason for<br>unsuccessful use | text | |

| Data file,<br>identifier patient | Notes | Variable<br>name | Variable<br>Iabel | Variable<br>Level | Nominal values |
|---|---|---|---|---|---|
| display id full | | | | | |
| data SAR | descriptive | n patadapt PA imp SAR <sup>52</sup> | Number of patient adapters | metric to be | o <b>1</b> |
| | | | PA used during implantation | reported as | o <b>2</b> |
| | | | | nominal | |
| | | n patadapt PA1B imp SAR <sup>53</sup> | Number of patient adapters | metric to be | o <b>1</b> |
| | | | PA1B used during | reported as | o <b>2</b> |
| | | | implantation | nominal | o |
| | | n patadapt PA1C imp SAR <sup>54</sup> | Number of patient adapters | metric to be | o <b>1</b> |
| | | | PA1C used during | reported as | o <b>2</b> |
| | | | implantation | nominal | |
| | | n patadapt PA2 imp SAR <sup>55</sup> | Number of patient adapters | metric to be | o <b>1</b> |
| | | | PA2 used during | reported as | o <b>2</b> |
| | | | implantation | nominal | |
| | | n patadapt nosuccess imp SAR <sup>56</sup> | Number patient adapters | metric to be | o <b>1</b> |
| | | | not successfully used during | reported as | o <b>2</b> |
| | | | implantation | nominal | |
| | | n patadapt problem imp SAR <sup>57</sup> | Number of used patient | metric to be | o <b>1</b> |
| | | | adapter with any problem | reported as | o <b>2</b> |
| | | | during implantation | nominal | |

<sup>&</sup>lt;sup>57</sup> Count QSPADPRB = "Yes, with Adverse Event" OR "Yes, without Adverse Event" per patient display id full



<sup>52</sup> Count DIPADMDL = "Patient adapter PA-1-B" OR "PA-1-C" OR "PA-2" per patient display id full

 $<sup>^{53}</sup>$  Count DIPADMDL = "Patient adapter PA-1-B" per patient display id full

<sup>&</sup>lt;sup>54</sup> Count DIPADMDL = "Patient adapter PA-1-C" per patient display id full

<sup>&</sup>lt;sup>55</sup> Count DIPADMDL = "Patient adapter PA-2" per patient display id full

<sup>&</sup>lt;sup>56</sup> Count QSPADAS = "used, but not successfully" per patient display id full

#### Accessory bag

| Data file, identifier<br>patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | Notes | | Variable<br>label | Variable<br>level | Nominal values |
|---|---|---|---|---|---|
| accessory log details (see Analysis Set and | no report | - | Usage of accessory bag | | o used successfully o used, but not successfully |
| Data Selection) | | | Did you notice any<br>problems related to<br>patient adapter | 1 | <ul><li>Yes, with Adverse Event</li><li>Yes, without Adverse Event</li><li>No problem detected</li></ul> |

| Data file, identifier<br>patient display id full &<br>SVTYP &<br>helpvar model &<br>DIPRGSNR | Notes | <br>Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|
| , 3 | case listing for<br>QSACCBAS = used, but not successfully OR<br>QSACCBPR = Yes, with Adverse Event OR<br>QSACCBPR = Yes, without Adverse Event<br>including programmer serial number<br>DIPRGSNR (see note before) | NEW: Accessory<br>bag: Please specify<br>reason for<br>unsuccessful use | text | |

| Data file,<br>identifier patient<br>display id full | Notes | Variable<br>name | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| data SAR | descriptive | n abag<br>imp SAR <sup>58</sup> | Number of accessory bags used during implantation | reported as | o1<br>o2<br> |
| | | n abag nosucccess<br>imp SAR <sup>59</sup> | , | reported as | o1<br>o2<br>o |
| | | 3 122 | Number of used accessory bag with any problem during implantation | reported as | o1<br>o2<br> |

<sup>60</sup> Count QSACCBPR = "Yes, with Adverse Event" OR "Yes, without Adverse Event" per patient display id full from the above selection of accessory log details



<sup>58</sup> Count non-missing QSACCBAS per patient display id full from the above selection of accessory log details

<sup>59</sup> Count QSACCBPR = "used, but not successfully" per patient display id full from the above selection of accessory log details

### 15.2. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4.

#### 15.3. Exclusion of Particular Information

See general definitions in chapter 5.5.

No data are excluded from the specified analysis set and variables.

## 15.4. Descriptive Analyses

For specification "Notes = descriptive", see general definitions in chapter 5.1.

## 15.5. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 16. Devices and Accessories - PHD & follow-up

#### CIP chapter 7.5 Further data of interest

General information

- · Implant type and model, all other implanted devices
- · Lead model and programmer software version

During implantation and follow-ups additional data on safety, performance and usability of the Renamic Neo system and accessories will be collected.

... Information on additionally used accessories or other implanted cardiac devices

### 16.1. Analysis Set and Data Selection

All analyses are performed for patients in the PHD and follow-up analysis set using a specific data selection after implantation<sup>61</sup>.

All analyses from chapter 15 Devices and Accessories - Implantation are repeated for these data. However, "implantation" will be replaced by and "PHD & follow-up".



<sup>&</sup>lt;sup>61</sup> analysis set PHD FUP SAR = Yes
Data selection for accessory log details with SVTYP ≠ implantation

## **Abbreviations**

ADE Adverse Device Effect

AE Adverse Event
AF Atrial Fibrillation

CDMS Clinical Data Management System

CI Confidence Interval

CIP Clinical Investigation Plan
CIR Clinical Investigation Report

CRF Case Report Form DD Device Deficiency

FU(P) Follow-up

PHD Pre-hospital discharge

SADE Serious Adverse Device Event

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAR Statistical Analysis Report

SOP Standard Operating Procedure

SD Standard Deviation

